CLINICAL TRIAL: NCT07196410
Title: A Phase I Study of KAN-004 in Patients With Immune-Related Diarrhea or Colitis
Brief Title: KAN-004 for Immune-Related Diarrhea or Colitis
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MP-02-2026-12952 (AE-KAN-004)
Record Dates: First submitted 2025-09-15; First posted 2025-09-29 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-08

CONDITIONS: Colitis; Diarrhea Caused by Antitumor Drugs
MeSH Terms: conditions — Colitis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants with steroid-naïve irColitis (Experimental): Participants with non-steroid refractory irColitis
  Interventions: Biological: KAN-004

INTERVENTIONS:
Biological: KAN-004 — Each dose of KAN-004 contains a consortium of bacteria isolated from the stool of healthy donors formulated as a powder in a capsule intended for oral administration

SUMMARY:
The goal of this clinical trial is to evaluate the safety and tolerability of KAN-004 in patients with immune-related colitis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of solid tumor treated with immune checkpoint inhibitor (≥1 cycle, ≤180 days since last cycle).
* Clinical diagnosis of irColitis (CTCAE >grade 2).
* Age ≥18 years
* Able to ingest capsules.
* Consent to provide blood and stool samples.
* Accessible for treatment and follow-up.
* Agreement to use highly effective contraception if of childbearing potential.

Exclusion Criteria:

* Prior/concurrent malignancy that could interfere with safety/efficacy assessment.
* Colostomy.
* Prior diagnosis of malabsorption.
* Untreated chronic hepatitis B or C.
* Solid organ transplant recipients.
* HIV-positive status.
* Pregnancy or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of KAN-004 | 6 weeks of treatment
  Proportion of participants with non-steroid refractory irColitis experiencing adverse events as measured by CTCAE v5.

CONTACTS AND LOCATIONS:
Overall Officials: Arielle Elkrief, MD, Principal Investigator — Centre Hospitalier de l'Universite de Montreal (CHUM)
Locations (1):
- Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec, Canada